CLINICAL TRIAL: NCT04758065
Title: Effectiveness of the Application of Radial Pressure Waves Together With a Manual Therapy Protocol and Therapeutic Exercise in the Treatment of Non-Specific Neck Pain: a Randomized Clinical Trial
Brief Title: Effectiveness of Radial Pressure Waves Therapy in the Treatment of Non-Specific Neck Pain (rPWT)
Acronym: rPWT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Pontificia Comillas (Other)
Responsible Party: Principal Investigator, Carlos López Moreno, Principal investigator, Universidad Pontificia Comillas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RPW-20/766-EC_X
Record Dates: First submitted 2021-02-08; First posted 2021-02-17 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Neck Pain
Keywords: Neck pain; Pain; Radial pressure waves; Elastography; Shear Wave; Physiotherapy; Exercise; Intervention
MeSH Terms: conditions — Neck Pain; Pain; Motor Activity | interventions — Exercise Therapy; Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: It is a randomized controlled clinical trial with parallel groups.
Masking Description: Blinding of investigators at study inclusion to randomization sequence, using sealed envelopes
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1-Goup: Control group (Active Comparator): Home-based cervical therapeutic exercise and manual therapy.
  Interventions: Other: Therapeutic Exercise and Manual Therapy
- 2-Group: Radial pressure waves Group (Experimental): Home-based cervical therapeutic exercise, manual therapy, and radial pressure waves.
  Interventions: Other: Radial pressure waves Therapy; Other: Therapeutic Exercise and Manual Therapy

INTERVENTIONS:
Other: Radial pressure waves Therapy — Combination of the usual physiotherapy treatment with the application of radial pressure waves compared with a control group in which only the usual treatment, in people with non-specific neck pain, will be applied.
  During the first month, the participants will perform 3 weekly sessions of home-based cervical therapeutic exercise and will come to the facilities, once a week, to get a manual therapy session based on the Maitland Concept (15 minutes of posteroanterior mobilizations in the restricted and/or painful vertebrae of the cervical and thoracic spine). Besides this participants of the experimental group will receive a radial pressure waves treatment sessión.
  Experimental Group: Home-based cervical therapeutic exercise, manual therapy, and radial pressure waves.
  Arms: 2-Group: Radial pressure waves Group
Other: Therapeutic Exercise and Manual Therapy — Combination of the usual physiotherapy treatment with the application of radial pressure waves compared with a control group in which only the usual treatment, in people with non-specific neck pain, will be applied.
  During the first month, the participants will perform 3 weekly sessions of home-based cervical therapeutic exercise and will come to the facilities, once a week, to get a manual therapy session based on the Maitland Concept (15 minutes of posteroanterior mobilizations in the restricted and/or painful vertebrae of the cervical and thoracic spine). Besides this participants of the experimental group will receive a radial pressure waves treatment sessión.
  Control Group: Home-based cervical therapeutic exercise and manual therapy.

SUMMARY:
The present study aims to know the effectiveness of radial pressure wave therapy in the treatment of people with nonspecific neck pain. The study hypothesis is that including radial pressure wave therapy in a protocol based on manual therapy and therapeutic exercise is more effective than the protocol alone for the treatment of nonspecific neck pain.

Participants will be randomly assigned into 2 groups, one will be applied only the manual therapy and exercise protocol and the other the same protocol, plus shock wave therapy. Data related to the pathology will be collected and compared between the two groups to determine which treatment is more effective.

DETAILED DESCRIPTION:
Nonspecific neck pain is one of the main reasons for outpatient physiotherapy consultation and, due to its multifactorial origin, there are numerous approaches without a consensus on the effectiveness of the different treatments. The most recent systematic reviews show significant evidence about the efficacy of the combination of Manual Therapy (MT) and exercise on pain, muscle elasticity, posture, and functionality in patients suffering from neck pain.

During muscle evaluation, it is common to find painful pressure points that are not spontaneously. These asymptomatic areas, painful when pressed, appear as areas with loss of elasticity, when evaluated with quantitative elastography (shear wave), which influences their contractile capacity and their ability to develop strength, together with the inhibition caused by the pain. The accumulation of cytotoxic and nociceptive substances, derived from the excess activity, could be the cause of the shortening of muscle fibers, so an increase in vascularity could help improve their drainage and normalize their elasticity and functionality.

Radial shock waves have been shown to be effective in angiogenesis, increasing vascularity and oxygen saturation of treated areas, so it could be a useful tool to help solve this problem.

This study aims to determine the effectiveness of radial shock waves to locate and treat the areas of loss of elasticity, found during muscle evaluation, combined with a MT and exercise protocol, compared to the manual therapy and exercise protocol itself. To do this, participants will be randomly assigned into 2 groups, one will be applied only the manual therapy and exercise protocol and the other the same protocol, plus shock wave therapy. The data collected will be compared between the two groups. An intention-to-treat statistical analysis will be performed.

Objective:

To determine the influence of the application of radial pressure waves together with the usual Physiotherapy treatment on the elasticity of muscle tissue, pain, the amplitude and harmony of cervical movements, strength, and quality of life in people with nonspecific neck pain

Methods:

The research will begin at the end of February 2021 and will be carried out in the biomechanics and movement analysis laboratory of the San Juan de Dios School of Nursing and Physiotherapy, Comillas Pontifical University, and at the Cimeg Madrid facilities.

A preliminary pilot study will be carried out with 10 volunteers with nonspecific neck pain, in order to calculate the sample size appropriate to the proposed objectives.

Participants will be randomly assigned using sealed envelopes to one of the two groups.

Group 1 will perform a conventional treatment protocol of physical therapy based on manual therapy and therapeutic exercise, for 4 weeks. Participants will go to the facilities, once a week, to get 1 session of manual therapy treatment, based on the Maitland Concept, on the cervical and thoracic spine. Besides this, they will perform 3 sessions a week of home-based cervical therapeutic exercise.

Group 2 will perform the same treatment protocol as Group 1, and in addition, will get a radial pressure waves session in the pressure sore spots, found in the muscle evaluation.

Muscle Elasticity, Pain Pressure Threshold, Cervical Pain, Active Range of Motion, the harmony of movement, Shoulder lift strength, Quality of life, Disability, and Kinesiophobia will be measured before and after treatment (at 4 weeks), at one month, and at three months after the start of the study. while demographic variables (Number of sore spots, Age, Sex, Dominance, Height, Weight, Body Mass Index (BMI), Educational level, Work Activity, and Sports Activity) will only be measured at the baseline.

.

ELIGIBILITY:
Inclusion Criteria:

* Non-Specific Neck Pain (NSNP)
* Age between 18 and 59 years,

Exclusion Criteria:

* Previous spine surgery.
* Neurological pathology.
* Rheumatoid arthritis.
* Fibromyalgia.
* Vertebral fractures or fissures.
* Radiculopathies.
* Neurogenic pain.
* History of cervical trauma.
* Congenital spinal anomalies.
* Wear a cardiac pacemaker.
* Currently receiving physiotherapy treatment in the same body area where the study is carried out.
* Currently being treated with anticoagulants or antiaggregants.
* Have an infectious or neoplastic nucleus close to the body area under study.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in Muscle Elasticity | Baseline, 4 weeks (after treatment), 1 month and 3 months after intervention commencement
  Using Shear Wave Elastography

SECONDARY OUTCOMES:
Change in Pain Pressure Threshold | Baseline, 4 weeks (after treatment), 1 month and 3 months after intervention commencement
  Using algometer
Change in Cervical Pain assessed by Visual Analog Scale for acute pain (Spanish version) | Baseline, 4 weeks (after treatment), 1 month and 3 months after intervention commencement
  Using Visual Analog Scale (VAS) for acute pain The VAS measures pain intensity with maximum reproducibility among observers. It consists of a horizontal line of 10 centimeters, at the ends of which are the extreme expressions of a symptom. In the left is the absence or less intensity and in the right the greater intensity. The patient is asked to mark on the line the point that indicates the intensity and it is measured with a millimeter ruler.
  Reliability (ICC = 0.96-0.98)
Change in Active Range of Motion | Baseline, 4 weeks (after treatment), 1 month and 3 months after intervention commencement
  Using the inertial sensor EBI 5.0 (ON) Biomedic. that provides information on the amplitude, speed, and acceleration of movements It is measured in degrees
Change in Jerk of cervical movements | Baseline, 4 weeks (after treatment), 1 month and 3 months after intervention commencement
  Using the inertial sensor EBI 5.0 (ON) Biomedic, that provides information on the amplitude, speed, and acceleration of movements.
  Jerk is a magnitude that measures the changes in acceleration during a movement, that is, the derivative of velocity with respect to time. For an angular movement, it is measured in (degrees/second^3)
Change in Shoulder lift strength | Baseline, 4 weeks (after treatment), 1 month and 3 months after intervention commencement
  Using Linear Encoder Chronojump The changes in the force that participants perform when lifting the shoulder will be measured, with the linear encoder in Newtons (N). Linear encoders are dynamometric devices that directly and continuously record the distance traveled and the movement time of a known external load, which therefore allows, through calculations, to obtain variables such as power and mechanical work, force or speed.
  Reliability: Pearson's correlation of all variables compared with the Biopac system (reference value) (≥0.94)
Change in the Quality of life assessed by the SF-12 questionnaire (Spanish version) | Baseline, 4 weeks (after treatment), 1 month and 3 months after intervention commencement
  Using SF-12 questionnaire. The SF-12 questionnaire (Spanish version) is a validated instrument to measure the Health-Related Quality of Life (HRQoL) of people. It consists of 12 items that collect measures on the functional and emotional state of the individual. When completing the questionnaire, the participant will obtain a value about their health between 1 and 5, where 1 is very good and 5 is bad.
  Reliability in all dimensions (Cronbach α ≥0.70)
Change in Disability assessed by the Neck disability index (NDI) questionnaire (Spanish version) | Baseline, 4 weeks (after treatment), 1 month and 3 months after intervention commencement
  Using Neck disability index (NDI) questionnaire. The Cervical Disability Index (NDI) is a 10-item questionnaire that measures disability related to neck pain reported by the patient. It offers 6 possible answers that represent 6 progressive levels of functional capacity and is scored from 0 to 5. The total score is expressed in percentage terms with respect to the maximum possible. The NDI is the most widely used questionnaire for neck pain. The NDI has been shown to be valid when compared to other measures of pain and disability.
  Reliability in all dimensions (Cronbach α = 0.944), intraclass correlation (0.98)
Change in Kinesiophobia assessed by the Tampa Scale for Kinesiophobia-11 (TSK-11) questionnaire (Spanish version) | Baseline, 4 weeks (after treatment), 1 month and 3 months after intervention commencement
  Using Tampa Scale for Kinesiophobia-11 (TSK-11) questionnaire (Spanish version).
  The Tampa Scale for Kinesiophobia (TSK) is one of the most widely used measures to assess pain-related fear in patients with pain.
  TSK is composed of 11 items, with a score range between 1 and 4, as follows: (1) Totally disagree, (2) Disagree, (3) Agree, (4) Totally agree. The total score of the scale range from 11- 44, where 11 means no kinesiophobia, 44 means severe kinesiophobia, and score ± 23 indicates there is kinesiophobia.
  Fiabilidad en todas las dimensiones (Cronbach α= 0.79), test-retest (ICC=0.81)
Number of sore spots | Baseline
  The variable "number of painful sore spots" in the assessed muscles, will be recorded in order to establish correlations with the dependent variables.
Age in years | Baseline
  The variable "age" of the participants will be recorded in order to establish correlations with the dependent variables.
Gender | Baseline
  The variable "gender" of the participants will be recorded in order to establish correlations with the dependent variables.
  Male/Female
Dominance | Baseline
  The variable "dominance" of the participants will be recorded in order to establish correlations with the dependent variables.
  Right/Left
Height in centimeters | Baseline
  The variable "Height" of the participants will be recorded, in centimeters, in order to establish correlations with the dependent variables.
Weight in kilograms | Baseline
  The variable "Weight" of the participants will be recorded, in kilograms, in order to establish correlations with the dependent variables.
Educational level | Baseline
  The variable "Educational level" of the participants will be recorded, using a shelf-completed registration document, in order to establish correlations with the dependent variables.
Work Activity | Baseline
  The variable "Work Activity" of the participants will be recorded, using a shelf-completed registration document, in order to establish correlations with the dependent variables.
Body Mass Index (BMI) | Baseline
  The variable "BMI" of the participants will be recorded, using a BMI calculator that combines the weight and height of the participants, in order to establish correlations with the dependent variables.
Sports Activity, assessed by Rapid Assessment of Physical Activity-1 (RAPA-1) test | Baseline
  The variable "Sports Activity" of the participants will be recorded, using the RAPA-1 test, in order to establish correlations with the dependent variables.
  RAPA-1 test is composed of 7 items related to the level of physical activity of the participants, with a score range between 1 and 7, as follows: (1) Sedentary (2-3) Not very active, (4-5) Moderately active, (6-7) active.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos López Moreno, MSc, Principal Investigator — San Juan de Dios School of Nursing and Phisiotherapy, Comillas Pontifical University
Locations (2):
- Spain (2):
  - San Juan de Dios School of Nursing and Phisiotherapy, Comillas Pontifical University, Ciempozuelos, Madrid
  - CIMEG Madrid, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Dissemination in biomedical research journals
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting January 2022
Access Criteria: Open Access

REFERENCES:
- [Background] Gerwin RD. Diagnosis of myofascial pain syndrome. Phys Med Rehabil Clin N Am. 2014 May;25(2):341-55. doi: 10.1016/j.pmr.2014.01.011. Epub 2014 Mar 18. PMID 24787337
- [Background] Hong CZ, Simons DG. Pathophysiologic and electrophysiologic mechanisms of myofascial trigger points. Arch Phys Med Rehabil. 1998 Jul;79(7):863-72. doi: 10.1016/s0003-9993(98)90371-9. PMID 9685106
- [Result] Madson TJ, Cieslak KR, Gay RE. Joint mobilization vs massage for chronic mechanical neck pain: a pilot study to assess recruitment strategies and estimate outcome measure variability. J Manipulative Physiol Ther. 2010 Nov-Dec;33(9):644-51. doi: 10.1016/j.jmpt.2010.08.008. Epub 2010 Oct 18. PMID 21109054
- [Result] Hidalgo B, Hall T, Bossert J, Dugeny A, Cagnie B, Pitance L. The efficacy of manual therapy and exercise for treating non-specific neck pain: A systematic review. J Back Musculoskelet Rehabil. 2017 Nov 6;30(6):1149-1169. doi: 10.3233/BMR-169615. PMID 28826164
- [Result] Ciubotariu A, Arendt-Nielsen L, Graven-Nielsen T. Localized muscle pain causes prolonged recovery after fatiguing isometric contractions. Exp Brain Res. 2007 Jul;181(1):147-58. doi: 10.1007/s00221-007-0913-4. Epub 2007 Mar 20. PMID 17372728
- [Result] Wang CJ, Ko JY, Chan YS, Weng LH, Hsu SL. Extracorporeal shockwave for chronic patellar tendinopathy. Am J Sports Med. 2007 Jun;35(6):972-8. doi: 10.1177/0363546506298109. Epub 2007 Feb 16. PMID 17307892
- [Result] Kraemer R, Sorg H, Forstmeier V, Knobloch K, Liodaki E, Stang FH, Mailaender P, Kisch T. Immediate Dose-Response Effect of High-Energy Versus Low-Energy Extracorporeal Shock Wave Therapy on Cutaneous Microcirculation. Ultrasound Med Biol. 2016 Dec;42(12):2975-2982. doi: 10.1016/j.ultrasmedbio.2016.08.010. Epub 2016 Sep 20. PMID 27662701
- [Result] Ballyns JJ, Turo D, Otto P, Shah JP, Hammond J, Gebreab T, Gerber LH, Sikdar S. Office-based elastographic technique for quantifying mechanical properties of skeletal muscle. J Ultrasound Med. 2012 Aug;31(8):1209-19. doi: 10.7863/jum.2012.31.8.1209. PMID 22837285
- [Result] Kozinc Z, Sarabon N. Shear-wave elastography for assessment of trapezius muscle stiffness: Reliability and association with low-level muscle activity. PLoS One. 2020 Jun 10;15(6):e0234359. doi: 10.1371/journal.pone.0234359. eCollection 2020. PMID 32520959
- See also: Tampa Scale for Kinesiophobia TSK-11 — https://ginvestigaciontmo.files.wordpress.com/2019/01/tsk-11-sv-spanish.pdf
- See also: NECK DISABILITY INDEX (NDI) Spanish Version — http://www.researchgate.net/publication/246617613_Validacion_de_una_version_espanola_del_Indice_de_Discapacidad_Cervical/link/59d92008a6fdcc2aad0d8ca7/download